CLINICAL TRIAL: NCT05711563
Title: Predicting and Monitoring Outcomes in Autoimmune Encephalitis
Acronym: POTA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Royal College of Surgeons, Ireland (Other)
Collaborators: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: 212573289
Record Dates: First submitted 2022-08-30; First posted 2023-02-03 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-01

CONDITIONS: Autoimmune Encephalitis
MeSH Terms: conditions — Autoimmune Diseases of the Nervous System | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — Serum and CSF
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Autoimmune Encephalitis (Ireland)
  Interventions: Other: Observational study
- Autoimmune Encephalitis (UK)
  Interventions: Other: Observational study
- Other neurological controls
  Interventions: Other: Observational study

INTERVENTIONS:
Other: Observational study — Observational study

SUMMARY:
Epilepsy is a disorder of the brain in which people have repeated seizures.

Autoimmune encephalitis (AE) is a rare cause of epilepsy. It is an inflammatory disease of the brain. This means that the body's own immune system attacks healthy brain tissue, just like it would if it were infected by a virus or a bacteria, by producing an army of proteins called 'antibodies' which go on to 'attack' healthy tissues.

Seizures in AE typically do not respond well to classic 'anti-seizure medications'. Instead, medications which suppress the immune system are used. These can have significant side-effects and some patients will still continue to have seizures or experience a recurrence of AE-related epilepsy despite treatment. It is difficult to accurately predict who will experience these outcomes.

This study aims to find ways of predicting and monitoring which people with AE are at greatest risk of these outcomes, so we can better direct them towards appropriate treatments. We will collect clinical information and samples of blood and cerebrospinal fluid (CSF, fluid surrounding the brain and spinal cord) from people with AE and 'control' participants with other neurological illnesses. Samples will be analysed for markers which may help predict or correlate with outcomes in AE and better understand this condition.

ELIGIBILITY:
Inclusion Criteria:

* AE participants over the age of 18 will be recruited if they meet the criteria for clinically probable or clinically definite Autoimmune Encephalitis as per Graus and colleagues 2016.
* Neurological Control participants undergoing lumbar puncture as part of clinical care for other, non-encephalitis disorders (e.g. for investigation of headache where meningitis or encephalitis is not detected, for investigation and treatment of idiopathic intracranial hypertension) in Beaumont hospital will be recruited.

Exclusion Criteria:

AE participants

* Under 18 years of age
* Participants without AE or those with a definitive alternate diagnosis for presentation.

Other neurological control participants will be excluded if they have a current or historic diagnosis of AE.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants with probable or definite autoimmune encephalitis will be recruited via the Oxford Autoimmune Neurology Group in the UK and Beaumont Hospital in Ireland.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Seizure frequency | 1-3 years
  >50% improvement in seizure frequency over time
Functional status | 1-3 years
  Modified Rankin score

SECONDARY OUTCOMES:
Cognitive ability | 1-3 years
  As measured by the Addenbrooke's Cognitive Examination.
Clinical status | 1-3 years
  As measured by the Clinical Assessment of severity in Autoimmune Encephalitis.
Mood/affect | 1-3 years
  Measured by the hospital anxiety and depression index
Quality of life | 1-3 years
  EQ-5D-5L (By EuroQOL, not an abbreviation)
Pain | 1-3 years
  Patient-Reported Outcomes Measurement Information System (PROMIS) Pain interference short form A
Fatigue | 1-3 years
  Fatigue Scale for Motor and Cognitive Funcitons
Fatigue | 1-3 years
  Modified Fatigue and Impact Scale
Sleep Quality | 1-3 years
  Pittsburgh Sleep Quality Index
Impulsivity | 1-3 years
  Barratt Impulsivity Index
Neuropsychiatric symptoms | 1-3 years
  Neuropsychiatric Inventory

OTHER OUTCOMES:
Other symptoms | 1-3 years
  Qualitiative analysis through semi-structured interview with participants and caregivers.

IPD SHARING:
Plan to Share IPD: Yes
Data or samples may (with consent) be shared in coded format with other ethically approved research studies, relating to disorders of the nervous system.
Access Criteria: Ethically approved studies which will process and dispose of data under the same regulations required by General Data Protection Regulation (GDPR) in Ireland and the European Union (EU).